CLINICAL TRIAL: NCT01115881
Title: Relationship Between Macular Thickness Measurement and Signal Strength Using Stratus Optical Coherence Tomography
Brief Title: Relationship Between Macular Thickness Measurement and Signal Strength in Optical Coherence Tomography
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: OCT-1
Record Dates: First submitted 2010-05-02; First posted 2010-05-04 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2010-01

CONDITIONS: Optical Tomography
Keywords: To examine the relationship between signal strength and macular thickness measured by stratus OCT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Signal strength is a parameter introduced in analysis software version 4.0.1, of the OCT stratus, that combines SNR and uniformity of the signal within a scan The scale of signal strength ranges from 1 to 10, with 1 representing poor image quality and 10 representing excellent image quality It has been showed that signal strength has a better image quality discriminating ability than SNR The operation manual recommends a minimum signal strength of 5 for macular thickness measurement There is no consensus on the level of signal strength above which should be considered to be good quality The inclusion Criteria for acceptable signal strength varies widely in the literature the purpose of our study is to examine the relationship between signal strength and macular thickness measured by stratus OCT

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects in this study other than refractive error, all included eyes had no concurrent ocular pathologic features BCVA of at least 20/30, and had spherical refractive error within the range of
* 4.00 D to 4.00 D

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ori Segal, M.D, Principal Investigator — Sackler school of medicine Tel-Aviv university
Locations (1):
- Meir medical center, Kfar Saba, Israel